CLINICAL TRIAL: NCT04676048
Title: Assessment of Safety and Preliminary Efficacy of ASC618 in Subjects With Severe and Moderately Severe Hemophilia A
Brief Title: ASC618 Gene Therapy in Hemophilia A Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ASC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-HA-001
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ASC618 (Experimental): Experimental Arm
  Interventions: Biological: ASC618

INTERVENTIONS:
Biological: ASC618 — ASC618 will be given as a single IV infusion

SUMMARY:
Currently, hemophilia A patients are managed with prophylactic or on-demand replacement therapy with recombinant FVIII or alternative therapeutics. The major challenges of current treatment regimens, such as the short half-life of hemophilia therapeutics with the need for frequent IV injections, encourage the current efforts for gene transfer therapy.

This study will evaluate the safety and preliminary efficacy of ASC618, an AAV vector encoding B-domain deleted codon-optimized human factor VIII under a synthetic liver-directed promoter

ELIGIBILITY:
Inclusion Criteria:

* Male ≥18 years of age
* Severe or moderately severe hemophilia A (FVIII activity ≤ 2 IU/dL) as evidenced by
* medical history
* Received FVIII prophylactic or on-demand replacement therapy for ≥ 150 accumulated
* days (exposure days)
* ≥12 bleeding episodes if receiving on-demand therapy over the preceding 12 months
* BMI ≤ 30
* Agree to use double-barrier contraceptive until at least 3 consecutive semen samples are negative after ASC-618 infusion

Exclusion Criteria:

* Pre-existing immunity to AAV8 vector as defined by AAV8 total antibodies and neutralizing antibodies qualified tests.
* Current inhibitors, or history of high titer FVIII inhibitors
* Presence of > Grade 2 liver fibrosis on elastography/Fibroscan or comparable imaging methodology
* History of chronic renal disease
* Active infection or any immunosuppressive disorder
* History of cardiac surgery and need anticoagulant therapy
* Any cardiovascular / genetic risk factors for thromboembolic disorders
* Evidence of active Hepatitis B, Hepatitis C, Human Immunodeficiency Virus (HIV)-1/2 or syphilis infection.
* Receipt of any vector or gene transfer agent
* Current antiviral therapy for hepatitis B or C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events, and serious AEs | 12 months post-infusion

SECONDARY OUTCOMES:
Changes in FVIII activity levels from baseline | 12 months post-infusion
Annualized FVIII consumption | 12 months post-infusion
Annualized bleeding rate (ABR) | 12 months post-infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No